CLINICAL TRIAL: NCT03484715
Title: Feasibility of a Physical Activity Programme Embedded Into the Daily Lives of Older Adults Living in Nursing Homes: a Randomised Controlled Pilot Feasibility Study
Brief Title: Feasibility of a Physical Activity Programme for Older Adults in Nursing Homes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Irish Research Council (Other)
Responsible Party: Principal Investigator, Eva Barrett, Postdoctoral Fellow, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GOIPD/2017/1301
Record Dates: First submitted 2018-03-06; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Old Age
Keywords: Physical Activity; Nursing Home; Feasibility; Older Adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomised controlled pilot feasibility study
Masking Description: As the primary aim of this study is to establish feasibility of the intervention and study processes, there will be no outcome assessor or participant blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Intervention (Experimental): Each participant in this arm will outline a small number of activity-related goals and will receive a 4 month personalised physical programme where additional physical activity will be incorporated into their daily routines. Nursing home staff will receive two educational sessions, which will provide them with the necessary skills to monitor participants physical activity programmes within the nursing home.
  Interventions: Behavioral: Physical Activity Intervention
- Usual Care Control (No Intervention): The participants in the control arm will receive usual care, which will be guided by current nursing and medical care plans.

INTERVENTIONS:
Behavioral: Physical Activity Intervention — A physical activity programme will be developed by the researcher for each participant. Integral to each physical activity programme will be a walking component (i.e. structured and gradual increases in daily walking time) and sit-to-stand exercises (i.e. a specified number of repeated rises from a chair). The rest of the physical activity programme will be tailored around each participant's specific functional goal and will be based on repeating particular functional activities. This programme will take place on 3 days per week in month 1, 4 days per week in month 2 and 3, and 5 days a week in month 4.
  Arms: Physical Activity Intervention

SUMMARY:
Older people living in nursing homes spend the majority of their time inactive. The current study has designed a physical activity intervention for older people living in nursing homes whereby the participants will incorporate more physical activity throughout their daily activities. Each participant's physical activity programme will be tailored to their physical abilities and to a pre-defined goal. The aim of this pilot feasibility study is to explore the feasibility and acceptability of this physical activity programme and to examine the preliminary effects of this on physical mobility and health-related quality of life, when compared to a usual care control group.

DETAILED DESCRIPTION:
Physical inactivity is a global health pandemic and is one of four leading contributors to premature mortality. Although there is evidence that physical activity improves short-term function and is safe among older adults of long-term care, the optimum contents of a physical activity programme or how best to implement it remain unclear. Few studies in nursing homes have attempted to increase physical activity levels by incorporating more usual activities into the resident's everyday routine. The proposed pilot feasibility study will implement a person-centred physical activity programme into the participant's daily routine, based on increasing duration and repetitions of everyday functions including walking and rising from a chair. It incorporates key constructs of social cognitive theory and is monitored by nursing home staff who will receive training and support.

Research questions:

This pilot feasibility study will have the following primary research questions:

1. Is the intervention feasible and acceptable to staff and participants?

   * Is the time commitment required for staff to monitor the intervention and participants to partake in the intervention feasible?
   * Are there any environmental barriers to completion of the intervention?
   * Is the content of the intervention acceptable to participants and staff?
   * Do the participants adhere to the intervention and what adherence issues arise?
2. Are the outcome measures feasible and acceptable to participants?

   * What is the required time and number of visits required to collect each outcome from participants?
   * Are the outcome measures acceptable to participants?
   * What is the level of missing data within the self-reported outcome measures?
3. What is the required sample size for a definitive randomised?

   * What is the baseline score and variability of the primary outcome measure among participants?
   * What is the estimated effect size and variance for the primary outcome measure?
   * What are the recruitment and attrition rates for nursing homes and participants? Do these rates differ between the intervention and control groups?

   The secondary research questions of the pilot study are:
4. What are the preliminary clinical outcomes and cost-effectiveness of the intervention compared to the control group?

   * What are the components of usual care for participants allocated to the control group?
   * What are the estimated outcomes of the intervention in comparison with the control group and are these sustained at 12 month follow-up?
   * What are the costs of the intervention in comparison to costs in the control group?
   * What is the feasibility of collecting health economic data (i.e. sources used and time taken)?

Design:

A randomised controlled pilot feasibility study, including a qualitative and economic component will be carried out. Two randomly selected nursing homes will take part in the study; participants (n=20) in one nursing home will receive the physical activity intervention and participants (n=20) in the other will receive usual care. In order to avoid contamination between intervention and control groups, randomisation will take place at nursing home level. The pilot feasibility study will not be an exact scale model of a definitive RCT, the difference being that outcome assessment will not be blinded as a full analysis of outcome data is not intended. However, the recruitment, randomisation, assessment and intervention conditions will be similar to a definitive RCT in order to answer the feasibility research questions. Quantitative outcome data will be collected in an unblinded manner from participants at T1 (baseline, pre-intervention), T2 (directly after completion of the intervention at 4 months) to examine the immediate intervention outcomes and T3 (12 months following the start of the intervention) to examine if the outcomes are sustained beyond intervention completion.

Qualitative component:

A qualitative descriptive approach will be taken for the qualitative component of the study. Qualitative data will be collected from participants and staff of the intervention group within 1 month following intervention completion and again with the participants at 7 months following intervention completion. Data will be collected via audio-recorded semi structured one-to-one interviews. The aim of the interviews with participants will be to explore the participant's experiences of receiving the intervention, the feasibility and acceptability of the intervention, the perceived effects of the intervention, including potential adverse effect, and issues around maintenance of the participants' physical activity over time, following intervention completion. The staff interviews will explore the staffs' role and experiences of being involved in the study, including their participation in the staff education sessions and the delivery of the physical activity programmes. Semi-structured qualitative interviews will be conducted with small subset of participants from the control group on two occasions. The first interviews will take place immediately following the recruitment and consent stage of the study, in order to maximise the feasibility data obtained for these study processes. The second interviews will take place upon completion of the 4 month intervention with the objective being to define and describe usual care.

Economic component:

A preliminary estimate of the costs and outcomes of the intervention relative to the usual care control will be assessed using a cost effectiveness analysis and cost utility analysis. Resource use associated with delivery of the physical activity intervention will be measured and costed. Resources used by participants over the course of the study will be recorded in both groups, for example health service usage, medication usage and private expenses relating to the intervention. Data collected from the primary outcome measure, the Timed Up and Go test, at each time point will be used alongside resource usage to provide the basis for the cost effectiveness analysis. For the cost utility analysis, effectiveness will be evaluated on the basis of the Quality Adjusted Life Year which will be estimated using the EuroQol 5 Dimensions 5 Levels instrument, assessed at baseline, 4 month and 12 month follow-up.

Statistical analysis:

SPSS Statistics (24.0 for Windows, Chicago, USA) will be use to analyse quantitative data. Demographical information in both groups will be tabulated and summarised. The effect of the intervention on clinical outcomes will be examined using suitable numerical and graphical summaries. The statistical analysis will serve primarily to provide an estimation of likely effect size and variance of effect size rather than statistical significance. Qualitative data will be analysed using NVivo (QSR International Pty Ltd. Version 11, 2015). Interviews will be transcribed verbatim and analysed using thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or over.
* Can speak and understand English.
* Resident in nursing home for at least 3 months.
* Able to rise from a chair with armrests (with or without a walking aid) and able to walk at least 10 metres (with or without a walking aid) independently or with minimal assistance.
* Approval of the resident's General Practitioner to participate.
* Cognitively capable of providing informed consent to participate, as judged by the key nurse caring for the participant.
* Cognitive function of a score of greater than 20 on the Mini Mental State Examination.

Exclusion Criteria:

* Admission to nursing home for respite or end-stage terminal care.
* A significant sensory impairment, physical impairment or illness that impairs their ability to participate.
* Uncontrolled cardiovascular, musculoskeletal or neurological disorders.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible nursing homes which agree to participate in study | Up to 2 months
  This will be expressed as a percentage of nursing homes which agree to participate in study out of the nursing homes which were invited to participle in study.
Proportion of eligible nursing home residents which agree to participate in study | Up to 1 month
  This will be expressed as a percentage of participants which agree to participate in study out of the participants which were invited to participle in study.
Time for recruitment of nursing homes | Up to 2 months
  This is be defined as time from initial contact with first nursing home to signing of final nursing home participation form and will be expressed as number weeks and days.
Time for recruitment of participants within nursing homes | Up to 1 month
  This is be defined as time from initial contact with first participant to signing of final participant consent form and will be expressed as number of weeks and days.
Retention rate of nursing homes at 4 month follow-up. | Assessed at 4 month follow-up.
  This is defined as percentage of nursing homes remaining in study at 4 month follow-up.
Retention rate of nursing homes at 12 month follow-up | Assessed at 12 month follow-up.
  This is defined as percentage of nursing homes remaining in the study at 12 month follow-up.
Retention rate of participants at 4 months | Assessed at 4 month follow-up
  This is defined as percentage of participants remaining in study at 4 month follow-up.
Retention rate of participants at 12 month follow-up | Assessed at 12 month follow-up.
  This is defined as percentage of participants remaining in the study at 12 month follow-up.
Adherence rate of participants to the intervention | Assessed at 4 month follow-up
  This will provide feasibility data. This will be expressed as the percentage of participants completing 75% of their physical activity programme according to the participant adherence sheets.

SECONDARY OUTCOMES:
Timed Up and Go Test | This will be assessed at baseline, directly after completion of the intervention at 4 months and at 12 months after the start of the intervention.
  This is a test of physical mobility and measures the time taken by an individual to stand up from a standard arm chair, walk a distance of 3 metres at a comfortable pace, turn, walk back to the chair, and sit down. Change in Timed Up and Go score will be measured in seconds.
Nottingham Health Profile | This will be assessed at baseline, directly after completion of the intervention at 4 months and at 12 months after the start of the intervention
  This provides a measure of health-related quality of life and change in Nottingham Health Profile score will be evaluated. The questionnaire measures self-perceived health across six domains: (i) sleep (ii) mobility (iii) energy (iv) pain (v) emotional reactions (vi) social isolation. Scores range from 0 to 1, with 0 indicating poor health and 1 indicating good health. There are no subscale scores to be reported.
10 Metre Walk Test | This will be assessed at baseline, directly after completion of the intervention at 4 months and at 12 months after the start of the intervention
  This is a measure of gait speed and the change in gait speed will be reported in seconds. The participant will walk 10 metres and the time is measured for the intermediate 6 metres to allow for acceleration and deceleration. The timer is started when the toes of the leading foot cross the 2-metre mark and stopped when the toes of the leading foot cross the 8-metre mark.
ICEpop CAPability measure for Older people (ICECAP-O) | This will be assessed at baseline, directly after completion of the intervention at 4 months and at 12 months after the start of the intervention.
  This provides a measure of capability-related quality of life and change in ICECAP-O score will be evaluated. The scale of this score ranges from 0 to 1, with 0 representing no capability and 1 representing full capability. There are no subscale scores to be reported.
Bangor Goal Setting Interview | This will be assessed at baseline, directly after completion of the intervention at 4 months and at 12 months after the start of the intervention
  In the intervention group only, the participant will rate their current performance and satisfaction with performance for their activity-based goal on a 1-10 Likert scale (where 1 means cannot do or am not doing successfully and 10 means can do and am doing very successfully). Change in scores will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Barrett, PhD, Principal Investigator — National Univeristy of Ireland, Galway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hallal PC, Andersen LB, Bull FC, Guthold R, Haskell W, Ekelund U; Lancet Physical Activity Series Working Group. Global physical activity levels: surveillance progress, pitfalls, and prospects. Lancet. 2012 Jul 21;380(9838):247-57. doi: 10.1016/S0140-6736(12)60646-1. PMID 22818937
- [Background] Crocker T, Forster A, Young J, Brown L, Ozer S, Smith J, Green J, Hardy J, Burns E, Glidewell E, Greenwood DC. Physical rehabilitation for older people in long-term care. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD004294. doi: 10.1002/14651858.CD004294.pub3. PMID 23450551
- [Background] Peri K, Kerse N, Robinson E, Parsons M, Parsons J, Latham N. Does functionally based activity make a difference to health status and mobility? A randomised controlled trial in residential care facilities (The Promoting Independent Living Study; PILS). Age Ageing. 2008 Jan;37(1):57-63. doi: 10.1093/ageing/afm135. Epub 2007 Oct 25. PMID 17965045
- [Background] Bandura A. Health promotion by social cognitive means. Health Educ Behav. 2004 Apr;31(2):143-64. doi: 10.1177/1090198104263660. PMID 15090118
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qualitative Research in Psychology. 3(2): 77-101, 2006.
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Holthe T, Thorsen K, Josephsson S. Occupational patterns of people with dementia in residential care: an ethnographic study. Scand J Occup Ther. 2007 Jun;14(2):96-107. doi: 10.1080/11038120600963796. PMID 17538854
- [Derived] Barrett E, Gillespie P, Newell J, Casey D. Feasibility of a physical activity programme embedded into the daily lives of older adults living in nursing homes: protocol for a randomised controlled pilot feasibility study. Trials. 2018 Aug 29;19(1):461. doi: 10.1186/s13063-018-2848-4. PMID 30157920